CLINICAL TRIAL: NCT01483885
Title: Comparison of the Analgesic Effects of Acupuncture and Modulated Electroanalgesia in Cold Induced Pain.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Assistant Professor at School of Physiotherapy, Universidade Federal do Piauí
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0208.0.045.000-11
Record Dates: First submitted 2011-11-23; First posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Cold Exposure
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- TENS 4Hz (Experimental)
  Interventions: Device: Transcutaneous Electric Nerve Stimulation
- Interferential Current 4Hz (Experimental)
  Interventions: Device: Interferential Current
- TENS (Placebo Comparator)
  Interventions: Device: Transcutaneous Electric Nerve Stimulation
- Interferential Current (Placebo Comparator)
  Interventions: Device: Interferential Current
- Manual Acupuncture (Experimental)
  Interventions: Procedure: Manual Acupuncture
- TENS 100 Hz (Experimental)
  Interventions: Device: Transcutaneous Electric Nerve Stimulation
- Interferential Current 100Hz (Experimental)
  Interventions: Device: Interferential Current

INTERVENTIONS:
Device: Transcutaneous Electric Nerve Stimulation — Tens at 4Hz and 100 Hz will be delivered using TENS stimulator (Ibramed/Neurodyn-São Paulo, Brazil)
  Arms: TENS; TENS 100 Hz; TENS 4Hz
Device: Interferential Current — Interferential Current (IC) at 4Hz and 100 Hz will be delivered using IC stimulator (Ibramed/Neurodyn-São Paulo, Brazil)
  Arms: Interferential Current; Interferential Current 100Hz; Interferential Current 4Hz
Procedure: Manual Acupuncture — Manual acupuncture will be delivered with sterile needles for each subject in the acupoint TA5 and CS6 localized in the dominant forearm.
  Arms: Manual Acupuncture

SUMMARY:
Physiotherapy offers a range of therapeutic modalities for pain management including Transcutaneous Electrical Nerve Stimulation (TENS), Interferential current (IC) and Acupuncture. The objective of this study was to investigate the hypoalgesic effect of TENS, CI and Acupuncture in a cold-induced pain model.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Subjects with no history of any kind of disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cold Pain threshold | 24 hours
  Cold pain threshold is recorded as the time from immersing the hand in the cold water to pain using a digital timer.

SECONDARY OUTCOMES:
Pain Tolerance threshold | 24 hours
  Cold Tolerance threshodl is recorded as the time from immersing the hand in the cold water to maximal pain tolerance using a digital timer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuad Ahmad Hazime, Parnaíba, Piauí, Brazil